CLINICAL TRIAL: NCT03456154
Title: Use of Botox Versus Conventional Treatment for Pain Decrease of Muscular Pain: a Randomized Controlled Trial
Brief Title: Botox vs Occlusal Splint for Masseter Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Maximiliano Sergio Cenci, PhD, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PPGO022
Record Dates: First submitted 2018-02-28; First posted 2018-03-07 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Pain, Face
MeSH Terms: conditions — Facial Pain | interventions — Occlusal Splints

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botox (Experimental): In this group patients will receive 3 injections of botox on each masseter (left and right), after randomization. This injection will be performed once, and the patient will be evaluated after 3 and 6 months after this day.
  Interventions: Drug: Botox Injectable Product
- Occlusal splint (Active Comparator): In this group patients will receive an occlusal splint, which will be manufactured after taking their full mouth impression. This appliance has to be worn everyday, for 6 months, at night.
  Interventions: Device: Occlusal splint

INTERVENTIONS:
Drug: Botox Injectable Product — 60u will be used at 3 sites of masseter muscle, on each side of the face
  Arms: Botox
Device: Occlusal splint — In this group patients will receive an occlusal splint which will be worn everyday for 6 months at night.
  Arms: Occlusal splint

SUMMARY:
This randomized clinical trial will compare the standard treatment (occlusal splint) and botox for the treatment of face muscular pain in adults. Fifty patients will be invited and selected, and allocated to the experimental group, according to the randomization sequence previously performed. For the splint group, a rigid splint will be worn by the patient every night. For the botox group, 60u of botox will be injected in 3 regions of the masseter muscle. Patients will be assessed before the experiment, 3 and 6 months after the beginning of the study. Oral health related quality of life, pain, and cervical neck position will be evaluated. Paired t-test and chi-square will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 70 years old;
* at least 20 teeth in the mouth;
* occlusal stability;
* presenting pain in face muscles.

Exclusion Criteria:

* Angle's Class III
* Kennedy's Class II or I removable partial denture wearer;
* Complete denture wearer;
* Individuals that have taken any anti inflammatory drugs in the last 3 months;
* Individuals with temporomandibular joint disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Masticatory muscle pain | baseline, 3 and 6 months
  VAS will be used to assess decrease of pain

SECONDARY OUTCOMES:
Oral health related quality of life | baseline, 3 and 6 months
  OHIP 14 questionnaire will be applied
Cervical Position | baseline, 3 and 6 months
  Modifications of cervical vertebral column position will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Pelotas, Pelotas, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Pires ALC, Galdino Santos L, Poletto-Neto V, Luz MS, Damian MF, Pereira-Cenci T. Evaluation of craniocervical posture after myofascial pain treatment in adults with bruxism: A randomized clinical trial. J Bodyw Mov Ther. 2024 Oct;40:1795-1801. doi: 10.1016/j.jbmt.2024.10.032. Epub 2024 Oct 16. PMID 39593526
- [Derived] Chisini LA, Pires ALC, Poletto-Neto V, Damian MF, Luz MS, Loomans B, Pereira-Cenci T. Occlusal splint or botulinum toxin-a for jaw muscle pain treatment in probable sleep bruxism: A randomized controlled trial. J Dent. 2024 Dec;151:105439. doi: 10.1016/j.jdent.2024.105439. Epub 2024 Nov 5. PMID 39510242